CLINICAL TRIAL: NCT04482946
Title: Dynamic Tests and Parameters to Predict Fluid Responsiveness After Off-pump Coronary Artery Bypass Grafting
Brief Title: Dynamic Tests and Parameters to Predict Fluid Responsiveness After OPCAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern State Medical University (Other)
Responsible Party: Principal Investigator, Mikhail Y. Kirov, Head of the anesthesiology and intensive care department, Northern State Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Dyn Test-and-Index
Record Dates: First submitted 2020-07-15; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Cardiac Surgery
Keywords: fluid responsiveness; dynamic tests; dynamic parameters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment of fluid responsiveness (Experimental): The positive end-expiratory pressure test (PEEP-test) consisted of a transient increase of PEEP from 5 to 20 cm H2O for 120 seconds. The PEEP-test was interrupted if MAP decreased below 55 mm Hg and/or pulse contour cardiac index (PCCI) decreased below 1.5 L/min/m2. Mini-fluid challenge test (mFCT) consisted of rapid infusion of crystalloids 1.5 mL/kg during 120 seconds. Thereafter, all patients received fluid challenge (standard fluid challenge test, sFCT). During the sFCT, patients received 7 mL/kg of crystalloids within 10 minutes. Investigators performed monitoring of mean arterial pressure (MAP), SVV and PPVPiCCO using femoral artery (PiCCO2). Investigators also assessed PVVNK using radial artery and Nihon Kohden patient monitor. HLI (Hamilton G-5, Switzerland) and PVI (Masimo, USA) were assessed non-invasively, using finger probes.
  Interventions: Diagnostic Test: Assessment of fluid responsiveness

INTERVENTIONS:
Diagnostic Test: Assessment of fluid responsiveness — The positive end-expiratory pressure test (PEEP-test) consisted of a transient increase of PEEP from 5 to 20 cm H2O for 120 seconds. The PEEP-test was interrupted if MAP decreased below 55 mm Hg and/or pulse contour cardiac index (PCCI) decreased below 1.5 L/min/m2. Mini-fluid challenge test (mFCT) consisted of rapid infusion of crystalloids 1.5 mL/kg during 120 seconds. Thereafter, all patients received fluid challenge (standard fluid challenge test, sFCT). During the sFCT, patients received 7 mL/kg of crystalloids within 10 minutes. Investigators performed monitoring of mean arterial pressure (MAP), SVV and PPVPiCCO using femoral artery (PiCCO2). Investigators also assessed PVVNK using radial artery and Nihon Kohden patient monitor. HLI (Hamilton G-5, Switzerland) and PVI (Masimo, USA) were assessed non-invasively, using finger probes.

SUMMARY:
Objective: To assess the predictive value of dynamic tests and parameters for evaluation of fluid responsiveness after off-pump coronary artery bypass grafting (OPCAB).

After arrival to ICU, all patients received positive end-expiratory pressure test (PEEP-test), mini-fluid challenge test (mFCT) and standard fluid challenge test (sFCT) to assess fluid responsiveness. In addition, investigators measured pulse pressure variation using two monitoring systems (PPVPiCCO and PPVNK), stroke volume variation (SVV), heart-lung interaction index (HLI) and plethysmogram variability index (PVI) before and after sFCT.

DETAILED DESCRIPTION:
All patients were intubated using the standard induction technique with sodium thiopental (4 mg/kg), fentanyl (2.5-3.0 mcg/kg) and pipecuronium bromide (0.1 mg/kg). Anaesthesia was maintained using sevoflurane (0.5-3.0 vol.% at the end of expiration) and fentanyl (2.0-4.0 mcg/kg/hr). Depth of anaesthesia was adjusted to maintain bispectral index (BIS) values between 40-60 (LifeScope, Nihon Kohden, Japan).

In all cases, preoxygenation with 80% O2 was provided during 3-5 minutes before anesthesia. After tracheal intubation, patients were ventilated using a protective volume-controlled mode (Dräger Primus, Germany) with tidal volume of 6-8 mL/kg of predicted body weight, flow of 1 L/min and positive end-expiratory pressure (PEEP) of 5 cm H2O. The value of FiO2 was set to at least 50% or higher to achieve intraoperative SpO2 above 95%. The respiratory rate was adjusted to maintain end-tidal CO2 values within 30-35 mm Hg.

All the patients were operated by the same team of surgeons using Acrobat SUV OM-9000S (Guidant, Santa Clara, USA) device for stabilization of the heart during revascularization.

After surgery, all patients were transferred to the postoperative cardiac ICU and sedated during 60 min with continuous infusion of propofol (2-4 mcg/kg/hr) to maintain BIS values within 60-70. Respiratory support in ICU was continued by a G5 ventilator (Hamilton Medical, Switzerland) using pressure controlled ventilation mode with parameters same as for intraoperative period.

Investigators provided invasive hemodynamic monitoring (PiCCO2, Pulsion Medical Systems, Germany; Nihon Kohden, MU-671RK, Japan) to all patients. After the initial stabilization of patient, investigators performed three dynamic tests in a consequent order. The positive end-expiratory pressure test (PEEP-test) consisted of a transient increase of PEEP from 5 to 20 cm H2O during 120 seconds. The PEEP-test was interrupted if mean arterial pressure (MAP) decreased below 55 mm Hg and/or pulse contour cardiac index (PCCI) decreased below 1.5 L/min/m2. Mini-fluid challenge test (mFCT) consisted of rapid infusion of crystalloids 1.5 mL/kg during 120 seconds. Thereafter, all patients received fluid challenge (standard fluid challenge test, sFCT). During the sFCT, patients received 7 mL/kg of crystalloids within 10 minutes. During PEEP-test and mFCT, investigators performed continuous monitoring of MAP, SVV, PPV and PCCI (PiCCO2). Investigators also measured SVV, PPVPiCCO, PVVNK (Nihon Kohden), HLI (Hamilton G-5, Switzerland) and PVI (Masimo, USA) before and after sFCT. In addition, investigators assessed cardiac index (CI), extravascular lung water index (EVLWI) and global end-diastolic volume index (GEDVI) using transpulmonary thermodilution (PiCCO2). During the study, investigators measured arterial blood gases and lactate concentration. The patients who demonstrated an increase in CI ≥ 15 % after sFCT were defined as fluid responders.10, 11 After the initial measurements, sedation was stopped, and the weaning from respiratory support was initiated. The weaning protocol included gradual decrease of inspiratory pressure and mandatory respiratory rate followed by spontaneous breathing trial after achieving pressure support of 8 cm H2O. After passing the 30-min spontaneous breathing trial, all the patients were extubated and received oxygen inhalation via facial mask.

In addition to hemodynamic and respiratory parameters, recorded the preoperative EuroScore II, duration of postoperative mechanical ventilation, length of ICU stay and fluid balance after OPCAB and on postoperative Day 1.

ELIGIBILITY:
Inclusion Criteria:

elective OPCAB

Exclusion Criteria:

morbid obesity with body mass index > 40 kg/m2 constant atrial fibrillation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Predictive value of dynamic tests | immediately postoperatively
  To assess if changes in mean arterial pressure, pulse pressure variation and stroke volume variation by more than 10% during the PEEP-test and mini fluid challenge test can predict the increment of the cardiac output on more than 15 % during standard fluid challenge test after off-pump coronary artery bypass grafting (OPCAB).

SECONDARY OUTCOMES:
Predictive value of dynamic parameters | immediately postoperatively
  To assess the ability of the decrement of Pulse pressure variation (measured by Nikhon), Heart-lung interaction index (HLI) and Pulse variability index (PVI) by more than 3% to predict the increment of the cardiac output on more than 15 % during standard fluid challenge test after off-pump coronary artery bypass grafting (OPCAB).

CONTACTS AND LOCATIONS:
Locations (1):
- City Hospital # 1 n.a. E.E. Volosevich, Arkhangelsk, Russia

IPD SHARING:
Plan to Share IPD: No